CLINICAL TRIAL: NCT03590275
Title: Observational Retrospective Study of Evaluation of Prognostic Factors in Advanced Pancreatic Cancer Patients Treated With FOLFIRINOX
Acronym: HOPE
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Alfredo Falcone, Prof. Alfredo Falcone, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: HOPE
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: pancreatic cancer; chemotherapy; FOLFIRINOX; prognostic
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: FOLFIRINOX — Patients treated with first-line FOLFIRINOX (oxaliplatin + irinotecan + lederfolin + 5-fluorouracil) as per clinical practice were included in the study

SUMMARY:
The aim of this study is to identify new prognostic factors in patients affected by advanced pancreatic carcinoma treated with first line chemotherapy with FOLFIRINOX regimen. Primary objective is the identification of clinical, laboratory and pathologic factors affecting overall survival of these patients.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* citologically or histologically confirmed pancreatic carcinoma
* disease stage III or IV according to the American Joint Committee on Cancer (AJCC) staging system
* access to clinical informations collected before first-line starting
* availability of objective response evaluation and survival data
* written informed consent

Exclusion Criteria:

* diagnosis of other neoplasia than pancreatic carcinoma
* treatment with drugs other than FOLFIRINOX
* treatment with experimental drugs in combination with FOLFIRINOX
* unavailability of clinical and pathological data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable advanced pancreatic carcinoma treated with FOLFIRINOX at the involved institutions between 2010 and 2017 will be included.
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 2 years
  Overall survival is defined as the time from study entry until death from any cause. Patients who are alive at the end of the study will be censored at that point.

SECONDARY OUTCOMES:
Progression-free survival | up to 2 years
  Progression-free survival is defined as time from study entry until progression of disease (according to RECIST 1.1) or death from any cause. Patients who are alive without having progressed at the end of the study will be censored at their last radiological assessment.
Response rate | up to 2 years
  Response rate is defined as the fraction of treated patients who achieve a response as defined according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria vers. 1.1.
Toxicity rate | up to 2 years
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing treatment-related adverse events as assessed by National Cancer Institute Common Toxicity Criteria (version 4.0), during chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Fornaro, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (7):
- Italy (7):
  - Oncologia ASL BI, Ponderano, Biella
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola, Forlì Cesena
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia FPO - IRCSS, Candiolo, Torino
  - ASL VCO, Ospedale Castelli Verbania, Verbania, Torino
  - A.O. Universitaria Pisana - Pisa (Pi) Oncologia Medica, Pisa
  - P.O. Molinette Oncologia 1, Torino
  - A.O. Ordine Mauriziano, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fornaro L, Leone F, Vienot A, Casadei-Gardini A, Vivaldi C, Lievre A, Lombardi P, De Luca E, Vernerey D, Sperti E, Musettini G, Satolli MA, Edeline J, Spadi R, Neuzillet C, Falcone A, Pasquini G, Clerico M, Passardi A, Buscaglia P, Meurisse A, Aglietta M, Brac C, Vasile E, Montagnani F. Validated Nomogram Predicting 6-Month Survival in Pancreatic Cancer Patients Receiving First-Line 5-Fluorouracil, Oxaliplatin, and Irinotecan. Clin Colorectal Cancer. 2019 Dec;18(4):e394-e401. doi: 10.1016/j.clcc.2019.08.004. Epub 2019 Sep 4. PMID 31564556